CLINICAL TRIAL: NCT07303712
Title: Liquid Biopsy for Hepatocellular Carcinoma Molecular Characterization and Assessment of Treatment Response After Y90 Radioembolization: A Pilot Study
Brief Title: Liquid Biopsy for Hepatocellular Carcinoma Molecular Characterization After Y90
Status: Recruiting | Type: Observational
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Sponsor
Other Study IDs: KIS0003ARG
Record Dates: First submitted 2025-03-17; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Circulating tumor cell (CTC); y90
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine if baseline liquid biopsy assays (CTC and cf-DNA) as well as single circulating tumor cell-DNA (sCTC DNA) dynamics in the early post-treatment period can predict subsequent treatment response to Y-90 radioembolization in patients with hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Study Aims and Objectives:

1. Assess the detection rate of CTC and cfDNA-based mutations and the distribution of molecular features of HCC prior to Y90 across BCLC A-C stages.
2. Determine CTC and cfDNA predictors at baseline that predict Y90 treatment response at 6-9 months.
3. Determine temporal changes in CTC and cfDNA mutations from baseline over 6-9 month course post Y90.
4. Determine if CTC mean distribution, sCTCDNA, and/or cfDNA mutational dynamic changes are predictive of treatment response at 6-9 months.
5. Assess radiomic and liquid biopsy signatures associated with outcome
6. Compare predictive outcome models using liquid biopsy data, imaging data, or a combination (multiomic data)

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18 years
2. HCC confirmed on imaging, BCLC stage 0, A, B, or C
3. Transarterial Y90 radioembolization approved by multidisciplinary tumor board -

Exclusion Criteria:

1. Not eligible for Y90 procedure
2. Prior surgery or ablation on indicated tumors
3. Patient unable to complete the follow up visits required for clinical care or research -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at VAPAHCS with HCC
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Circulating Tumor Cell (CTC) | Baseline, 1 month post treatment, 3 months post treatment, and 6 months post treatment
  blood samples
CTA imaging | Baseline, 3 months post treatment, 6 months post treatment
  imaging of liver tumor

CONTACTS AND LOCATIONS:
Overall Officials: Sirish Kishore, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT07303712/ICF_000.pdf